CLINICAL TRIAL: NCT01076140
Title: Comparative Blood Pressure Effects of Nebivolol Versus Lisinopril in Patients With New Onset or Exacerbated Hypertension Induced by Bevacizumab: a Crossover Study
Brief Title: Blood Pressure Effects of Nebivolol Versus Lisinopril in New Onset or Worsening Hypertension Induced by Bevacizumab
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Zachery Somers, PharmD, University of Mississippi Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0222
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Hypertension
Keywords: Hypertension as a result of bevacizumab therapy
MeSH Terms: conditions — Hypertension | interventions — Nebivolol; Lisinopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebivolol (Active Comparator): Nebivolol 5 mg daily for 2 weeks, then 5 or 10 mg daily for 2 weeks
  Interventions: Drug: Nebivolol
- Lisinopril (Active Comparator): 20 mg once daily for 2 weeks, then 20 or 40 mg once daily for 2 weeks
  Interventions: Drug: Lisinopril

INTERVENTIONS:
Drug: Nebivolol — Nebivolol 5 or 10 mg tablets daily for 4 weeks. Lisinopril 20 or 40 mg daily for 4 weeks
  Arms: Nebivolol
Drug: Lisinopril — Nebivolol 5 or 10 mg tablets daily for 4 weeks. Lisinopril 20 or 40 mg daily for 4 weeks
  Arms: Lisinopril

SUMMARY:
The purpose of this study is to directly compare the blood pressure (hypertension) reduction effects of lisinopril and nebivolol in patients who develop new onset or worsening hypertension while treated with bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients currently treated at the University of Mississippi Medical Center Oncology Clinic
* Patient is being treated with bevacizumab either alone or in combination with other agents for cancer
* Patient blood pressure is >140 mmHg (systolic) or > 90 mmHg (diastolic), either treated or untreated with medications for hypertension
* Patients may be currently on medications for hypertension (other than Beta blocker, ACEI, or ARB); these will be continued at the same dose throughout the study
* Patients should be > 18 years of age
* Patients receiving bevacizumab therapy approximately every 2 weeks

Exclusion Criteria:

* History of ACEI or ARB induced angioedema or idiopathic/hereditary angioedema
* Patient currently treated with a Beta blocker, ACEI, or ARB or have a history of intolerance to a medication in any of these classes
* Hyperkalemia, defined as a potassium value of >5 mEq/L
* Pregnancy or breastfeeding
* Severe renal impairment (eGFR <30 mL/min)
* Moderate hepatic impairment as identified by physician
* Currently taking CYP2D6 inducers (rifampin, carbamazepine or dexamethasone) or inhibitors (bupropion, fluoxetine, paroxetine, duloxetine, etc.)
* History of clinically significant EKG abnormality which would contraindicate beta blocker use
* Recent stroke (<6 months)
* Recent myocardial infarction (<6 months)
* Congestive heart failure
* Severe asthma or COPD
* Diagnosed obstructive sleep apnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2011-01 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the study will be changes in sitting systolic and diastolic blood pressure at the crossover and final visits. | 8 weeks
  Patients will be treated with both nebivolol or lisinopril for a period of 4 weeks, and then crossover to the opposite medication for an additional 4 weeks.

SECONDARY OUTCOMES:
The secondary endpoint of the study will be changes in heart rate at the end of the crossover and final visits. | 8 weeks
  Patients will be treated with both nebivolol or lisinopril for a period of 4 weeks, and then crossover to the opposite medication for an additional 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States